CLINICAL TRIAL: NCT03030768
Title: Pilot of an mHealth-enhanced, Safer Conception Intervention to Reduce HIV-1 Risk Among Kenyan HIV-1 Serodiscordant Couples
Brief Title: Safer Conception Intervention for HIV-1 Serodiscordant Couples
Acronym: SCIP
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Renee Heffron, Assistant Professor, University of Washington
Other Study IDs: STUDY00002068; R00HD076679 (NIH); R21TW009908 (NIH)
Record Dates: First submitted 2017-01-12; First posted 2017-01-25 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: HIV Seropositivity; Pregnancy, High-Risk
Keywords: Pre-Exposure Prophylaxis; Fertility; mHealth; Pregnancy
MeSH Terms: conditions — HIV Seropositivity | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-1 serodiscordant couples: Couples where one partner is HIV-1 infected and the other is uninfected, who will receive counseling on timed condomless sex, ART and PrEP adherence. The study intervention focuses on ART use by the HIV-1 infected partner, PrEP (Truvada) use by the HIV-1 uninfected partner, and timed condomless sex during the peri-conception period.
  Interventions: Drug: PrEP; Behavioral: Counseling on timed condomless sex, ART and PrEP adherence

INTERVENTIONS:
Drug: PrEP — An integrated, phased safer conception intervention that focuses on ART use by the HIV-1 infected partner, PrEP use by the HIV-1 uninfected partner, and timed condomless sex during the peri-conception period.
  Other Names: Truvada
Behavioral: Counseling on timed condomless sex, ART and PrEP adherence — An integrated, phased safer conception intervention that focuses on ART use by the HIV-1 infected partner, PrEP use by the HIV-1 uninfected partner, and timed condomless sex

SUMMARY:
The greatest burden of the HIV-1 epidemic lies in sub-Saharan Africa, where a substantial proportion of infections occur in long-term heterosexual HIV-1 serodiscordant partnerships. Such couples face a difficult dilemma when considering their desire to have children: forego condom use, attempt to conceive and risk HIV-1 transmission or continue condom use and relinquish their childbearing desires. Based on evidence from rigorous clinical trials demonstrating the strong efficacy of individual interventions for HIV-1 prevention and formative work with HIV-1 serodiscordant couples and clinicians with expertise in HIV-1 prevention and reproductive health in the Kenyan context, this study pilots a safer conception intervention that focuses on antiretrovirals (as antiretroviral therapy [ART] taken by the HIV-1 infected partner and pre-exposure prophylaxis [PrEP] taken by the HIV-1 uninfected partner) and timed condomless sex. Additional strategies for couples include diagnosis and treatment of STIs and male circumcision.

mHealth tools, including SMS and mobile applications are novel and very popular among Kenyans to ease the burden of addressing health problems. This safer conception intervention incorporates mHealth tools to improve couples' experiences tracking fertility indicators and communicating with providers about their readiness to practice safer conception. SMS surveys to collect daily information from women about their fertility signs and SMS messages are used to reinforce HIV-1 prevention, including condom use for couples during periods that do not have a high likelihood of fertility. An in-clinic mobile application is used to improve clinician-patient counseling and assessments of couple readiness to practice safer conception. To inform future engagement of mHealth tools, the investigators will prospectively evaluate clinician and patient experiences using SMS surveys and the tablet application. Couples with immediate fertility intentions will be followed longitudinally, allowing careful tracking of pregnancy and HIV-1 incidence. The study takes place in Thika, Kenya.

DETAILED DESCRIPTION:
Overall Design This is an open-label, prospective cohort pilot study of HIV-1 serodiscordant couples with immediate fertility desires. The overall goal is to determine uptake and sustained use of safer conception strategies, strategies for HIV-1 risk reduction during periods when couples attempt to conceive a child. The study offers PrEP (daily oral TDF or FTC/TDF) to the HIV-1 uninfected member of the couple, ART to the HIV-1 infected member of the couple, teach women about tracking fertility indicators and predicting upcoming periods of peak fertility, and work with couples to establish their readiness to practice timed condomless sex. mHealth tools will be integrated to capture fertility indicators, sexual behavior, improve patient-provider communication, and remind couples about their upcoming periods with peak fertility. The investigators will conduct mixed-methods work to understand couples experiences practicing safer conception and couples and providers experiences using the mHealth tools.

AIMS

1. To determine uptake (and adherence, when applicable) of each component of an integrated safer conception intervention among HIV-1 serodiscordant couples, including:

   1. Use of PrEP by the HIV-1 uninfected partner
   2. Use of ART by the HIV-1 infected partner
   3. Menstrual cycle monitoring
   4. Patterns of condom use
   5. STI treatment
   6. Medical male circumcision, and
   7. Vaginal self-insemination
2. To determine rates of pregnancy and HIV-1 incidence among HIV-1 serodiscordant couples participating in a safer conception intervention pilot
3. To determine which fertility indicators - including onset of menses, basal body temperature, vaginal mucus characteristics, results from luteinizing hormone tests - are most feasible for Kenyan women in HIV-1 serodiscordant partnerships to monitor via SMS
4. To obtain user feedback about mHealth tools designed to improve patient experience with safer conception including:

   1. Women's experiences tracking fertility signs through SMS and
   2. Couples' and provider's experiences using a clinic-based tablet application that encompasses clinical, laboratory and fertility data to improve patient-provider communication about safer conception readiness
   3. Women and men's experiences receiving SMS messages with personalized safer conception reminders
5. To assess participant experiences with an mHealth-enhanced safer conception intervention

Study procedures:

Clinic visits will take place at screening and enrollment, monthly prior to pregnancy and quarterly during pregnancy, for up to 12 months or the end of pregnancy, whichever comes later. Couples will move from a preparatory period into a peri-conception period once they decide to practice timed condomless sex, based on discussions with study clinicians and counselors. They will move from peri-conception to pregnancy once pregnancy occurs or from peri-conception to study exit if pregnancy does not occur within 12 months of study enrollment. During the preparatory and peri-conception periods, women will receive daily SMS surveys.

Screening:

At screening, both members of couples will undergo HIV-1 testing to verify HIV-1 serodiscordancy and women will have a pregnancy test. Demographic, behavioral and medical information will be collected, along with additional laboratory results to establish eligibility (for HIV-1 uninfected partners - serum creatinine, hepatitis B surface antigen). Couples' fertility desires will be assessed and medical history will include information about current use of contraceptives and menstrual cycle regularity.

Enrollment:

At enrollment, members of couples will separately complete interviewer-administered questionnaires to assess their pre-intervention knowledge, perceptions of, and barriers to safer conception strategies and gather data on their demographic and medical characteristics, sexual behavior and any current contraception and/or antiretroviral use. Both partners will undergo diagnostic testing and treatment of genital infections, including gonorrhea, chlamydia, trichomonas, and bacterial vaginosis (BV, if there are symptoms). HIV-1 uninfected partners will be re-tested to verify their HIV-1 status and assessed for acute HIV-1 infection. Women will be tested for pregnancy. HIV-1 infected partners will have specimen collected for CD4 and plasma viral load quantification. Physical exams will be conducted for both partners. Social harm will also be assessed in a culturally appropriate manner and captured on validated case report forms. Safer conception behavioral counseling will be in addition to couples counseling for HIV-1 prevention that fosters an understanding of HIV-1 serodiscordancy and negotiation of safer sex.

Daily SMS surveys:

The day after enrollment, women will begin to receive daily SMS surveys to assess fertility signs and sexual behavior.

Follow up visits:

Participants will complete follow up visits to track their compliance with the intervention strategies and study procedures. Participants will be scheduled for monthly study visits during the preparatory and peri-conception periods and quarterly during pregnancy. Participants can move from the preparatory period to peri-conception based on their own desires and counseling from a clinician.

Exit:

Following the end of pregnancy or 12 months after study enrollment (whichever is later), couples will be exited from the study. At study exit, couples will be counseled about their current fertility goals (which may have changed throughout the course of follow up, especially for couples who become pregnant and have a child during the study period) and offered contraception and referrals for ongoing services, as appropriate.

Qualitative interviews:

To gain a deeper understanding of how participants perceive the integrated safer conception intervention and the mHealth components that are part of the intervention, we will conduct in-depth interviews with up to 40 couples. Interview topics will include: identification of factors influencing individuals' preferences for safer conception strategies, their experience with safer conception strategies, and their intentions for continued use of these strategies should they desire pregnancy again and user satisfaction with the mHealth tools and suggestions for improvement.

ELIGIBILITY:
Inclusion Criteria:

* Couples

  * Immediate fertility intention
  * Sexually active (defined as having had vaginal intercourse at least 6 times in the previous three months)
  * Willing to enter the study as a couple and intending to remain as a couple for the next 12 months

For HIV-1 infected members of the couple (index participants)

* Able and willing to provide written informed consent
* HIV-1 infected based on positive rapid HIV-1 tests, according to national algorithm
* Not currently pregnant or breastfeeding
* No use of injectable contraception for the past 3 months
* Not currently enrolled in an HIV-1 treatment study
* No clear indication of infertility or subfertility, as determined by medical history
* Own a mobile phone for personal use, which operates on a telecom provider supported by the study SMS platform and is distinct from the mobile phone owned by the HIV-1 uninfected partner
* Know how to send and receive SMS
* Have regular access to electricity or an alternative means for charging a cell phone Literate in English, Kiswahili or Kikuyu

For HIV-1 uninfected members of the couple (partner participants)

* Able and willing to provide written informed consent
* HIV-1 uninfected based on negative HIV-1 rapid tests, both at study screening and at the enrollment visit
* Adequate renal function, defined by normal creatinine levels and estimated creatinine clearance ≥60 mL/min
* Not infected with hepatitis B virus, as determined by a negative hepatitis B surface antigen test
* Not currently pregnant or breastfeeding
* No use of injectable contraception for the past 3 months
* Not currently enrolled in an HIV-1 prevention clinical trial
* Enrollment of individuals with active and serious infections or active clinically significant medical problems will be at the discretion of the site investigator
* No clear indication of infertility or subfertility, as determined by medical history
* Own a mobile phone for personal use, which operates on a telecom provider supported by the study SMS platform and is distinct from the mobile phone owned by the HIV-1 infected partner
* Know how to send and receive SMS
* Have regular access to electricity or an alternative means for charging a cell phone
* Literate in English, Kiswahili or Kikuyu

For study clinicians and counselors

• Active involvement in safer conception counseling for couples and use of the tablet application during counseling sessions

Exclusion Criteria:

* For couples

  * Participated in the Partners PrEP Study or the Partners Demonstration Project For HIV-1 infected members of the couple (index participants)
  * Currently pregnant or breastfeeding
  * Used an injectable contraception in the past 3 months
  * Currently enrolled in an HIV-1 treatment study
  * Has a clear indication of infertility or sub-fertility, as determined by medical history

For HIV-1 uninfected members of the couple (partner participants):

* Infected with hepatitis B virus, as determined by a positive hepatitis B surface antigen test
* Currently pregnant or breastfeeding
* Used an injectable contraception in the past 3 months
* Currently enrolled in an HIV-1 prevention clinical trial
* Has a clear indication of infertility or subfertility, as determined by medical history
* Enrollment of individuals with active and serious infections or active clinically significant medical problems will be at the discretion of the site investigator

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Heterosexual HIV-1 serodiscordant couples in Thika, Kenya with immediate fertility desires, who did not participate in a previous study "Partners PrEP Study or the Partners Demonstration Project" at the site, and study clinicians and counselors delivering the intervention.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-02; Primary Completion 2018-05 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Pregnancy incidence - rate of pregnancy that occurs per 12 months | 12 months post enrollment
  Rate of pregnancy that occur without HIV-1 transmission to the uninfected partner

SECONDARY OUTCOMES:
HIV-1 incidence - rate of new HIV infections that occur per 12 months | 12 months post enrollment
  Rate of new HIV-1 infections among couples

OTHER OUTCOMES:
User feedback about mHealth tools designed to improve patient experience with safer conception | 12 months post enrollment
  Women's experiences tracking fertility signs through SMS. Couples' and provider's experiences using a clinic-based mobile application that encompasses clinical, laboratory and fertility data to improve patient-provider communication about safer conception readiness

CONTACTS AND LOCATIONS:
Overall Officials: Renee Heffron, PhD, Study Chair — University of Washington
Locations (2):
- University of Washington, Coordinating Center, Seattle, Washington, United States
- Partners in Health, Research and Development, Thika, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all outcome measures will be made available after study completion

REFERENCES:
- [Background] Heffron R, Ngure K, Mugo N, Celum C, Kurth A, Curran K, Baeten JM. Willingness of Kenyan HIV-1 serodiscordant couples to use antiretroviral-based HIV-1 prevention strategies. J Acquir Immune Defic Syndr. 2012 Sep 1;61(1):116-9. doi: 10.1097/QAI.0b013e31825da73f. PMID 22595872
- [Background] Ngure K, Baeten JM, Mugo N, Curran K, Vusha S, Heffron R, Celum C, Shell-Duncan B. My intention was a child but I was very afraid: fertility intentions and HIV risk perceptions among HIV-serodiscordant couples experiencing pregnancy in Kenya. AIDS Care. 2014;26(10):1283-7. doi: 10.1080/09540121.2014.911808. Epub 2014 Apr 29. PMID 24779445
- [Background] Guidance on Couples HIV Testing and Counselling Including Antiretroviral Therapy for Treatment and Prevention in Serodiscordant Couples: Recommendations for a Public Health Approach. Geneva: World Health Organization; 2012 Apr. Available from http://www.ncbi.nlm.nih.gov/books/NBK138278/ PMID 23700649
- [Background] Irungu EM, Heffron R, Mugo N, Ngure K, Katabira E, Bulya N, Bukusi E, Odoyo J, Asiimwe S, Tindimwebwa E, Celum C, Baeten JM; Partners Demonstration Project Team. Use of a risk scoring tool to identify higher-risk HIV-1 serodiscordant couples for an antiretroviral-based HIV-1 prevention intervention. BMC Infect Dis. 2016 Oct 17;16(1):571. doi: 10.1186/s12879-016-1899-y. PMID 27751179
- [Background] Mugo NR, Hong T, Celum C, Donnell D, Bukusi EA, John-Stewart G, Wangisi J, Were E, Heffron R, Matthews LT, Morrison S, Ngure K, Baeten JM; Partners PrEP Study Team. Pregnancy incidence and outcomes among women receiving preexposure prophylaxis for HIV prevention: a randomized clinical trial. JAMA. 2014 Jul 23-30;312(4):362-71. doi: 10.1001/jama.2014.8735. PMID 25038355
- [Background] Baeten JM, Donnell D, Ndase P, Mugo NR, Campbell JD, Wangisi J, Tappero JW, Bukusi EA, Cohen CR, Katabira E, Ronald A, Tumwesigye E, Were E, Fife KH, Kiarie J, Farquhar C, John-Stewart G, Kakia A, Odoyo J, Mucunguzi A, Nakku-Joloba E, Twesigye R, Ngure K, Apaka C, Tamooh H, Gabona F, Mujugira A, Panteleeff D, Thomas KK, Kidoguchi L, Krows M, Revall J, Morrison S, Haugen H, Emmanuel-Ogier M, Ondrejcek L, Coombs RW, Frenkel L, Hendrix C, Bumpus NN, Bangsberg D, Haberer JE, Stevens WS, Lingappa JR, Celum C; Partners PrEP Study Team. Antiretroviral prophylaxis for HIV prevention in heterosexual men and women. N Engl J Med. 2012 Aug 2;367(5):399-410. doi: 10.1056/NEJMoa1108524. Epub 2012 Jul 11. PMID 22784037
- [Background] Mugo NR, Heffron R, Donnell D, Wald A, Were EO, Rees H, Celum C, Kiarie JN, Cohen CR, Kayintekore K, Baeten JM; Partners in Prevention HSV/HIV Transmission Study Team. Increased risk of HIV-1 transmission in pregnancy: a prospective study among African HIV-1-serodiscordant couples. AIDS. 2011 Sep 24;25(15):1887-95. doi: 10.1097/QAD.0b013e32834a9338. PMID 21785321
- [Background] Baeten JM, Heffron R, Kidoguchi L, Mugo NR, Katabira E, Bukusi EA, Asiimwe S, Haberer JE, Morton J, Ngure K, Bulya N, Odoyo J, Tindimwebwa E, Hendrix C, Marzinke MA, Ware NC, Wyatt MA, Morrison S, Haugen H, Mujugira A, Donnell D, Celum C; Partners Demonstration Project Team. Integrated Delivery of Antiretroviral Treatment and Pre-exposure Prophylaxis to HIV-1-Serodiscordant Couples: A Prospective Implementation Study in Kenya and Uganda. PLoS Med. 2016 Aug 23;13(8):e1002099. doi: 10.1371/journal.pmed.1002099. eCollection 2016 Aug. PMID 27552090
- [Background] Matthews LT, Heffron R, Mugo NR, Cohen CR, Hendrix CW, Celum C, Bangsberg DR, Baeten JM; Partners PrEP Study Team. High medication adherence during periconception periods among HIV-1-uninfected women participating in a clinical trial of antiretroviral pre-exposure prophylaxis. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):91-7. doi: 10.1097/QAI.0000000000000246. PMID 25118795
- [Background] Heffron R, Pintye J, Matthews LT, Weber S, Mugo N. PrEP as Peri-conception HIV Prevention for Women and Men. Curr HIV/AIDS Rep. 2016 Jun;13(3):131-9. doi: 10.1007/s11904-016-0312-1. PMID 26993627
- [Derived] Heffron R, Ngure K, Velloza J, Kiptinness C, Quame-Amalgo J, Oluch L, Thuo N, Njoroge J, Momanyi R, Gakuo S, Mbugua S, Morrison S, Haugen H, Chohan B, Celum C, Baeten JM, Mugo N. Implementation of a comprehensive safer conception intervention for HIV-serodiscordant couples in Kenya: uptake, use and effectiveness. J Int AIDS Soc. 2019 Apr;22(4):e25261. doi: 10.1002/jia2.25261. PMID 30957420